CLINICAL TRIAL: NCT01847963
Title: Standardization and Clinical Evaluation of Siddha Formulations for Urolithiasis /Kalladaippu.
Brief Title: A Clinical Study to Evaluate the Efficacy of Two Siddha Drugs Sindhuvallathy Mezhugu and Kalladaippu Kudineer for Kidney Stones
Acronym: SVMKK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Collaborators: University Grants Commission (Other); Tamilnadu Dr MGR Mecical University research council (Unknown)
Responsible Party: Principal Investigator, Dr. K. Rajalakshmi, Assistant professor, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGR-10-KR- 1301; BCR - 2043 (Other Grant/Funding Number: UGC minor project F.no 41-1432-2011)
Record Dates: First submitted 2013-04-23; First posted 2013-05-07 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Kalladaippu Kudineer; Siddha; Sindhuvallathy; Kidney stones
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sindhuvallathy mezhugu (Experimental): Sindhuvallathy mezhugu (SVM) 500 mg Twice daily per Oral 45 days duration
  Interventions: Drug: Sindhuvallathy mezhugu ( SVM)
- Kalladaippu Kudineer (Experimental): Kalladaippu Kudineer (KK) 130 ml decoction Twice daily Per oral 45 days Duration
  Interventions: Drug: Kalladaippu Kudineer (KK) -
- Sindhuvallathy + Kalladaippu Kudineer (Experimental): Sindhuvallathy mezhu -500 mg capsules twice daily + Kalladaippu kudineer -130 ml decoction twice daily-per oral for 45 days.
  Interventions: Drug: Sindhuvallathy mezhugu ( SVM); Drug: Kalladaippu Kudineer (KK) -

INTERVENTIONS:
Drug: Sindhuvallathy mezhugu ( SVM) — 500 mg capsules per oral twice daily for 45 days a Siddha classical literature preparation
  Arms: Sindhuvallathy + Kalladaippu Kudineer; Sindhuvallathy mezhugu
Drug: Kalladaippu Kudineer (KK) - — 130 ml decoction twice daily-per oral for 45 days, a Siddha classical literature preparation
  Other Names: Sirupeelai kudineer
  Arms: Kalladaippu Kudineer; Sindhuvallathy + Kalladaippu Kudineer

SUMMARY:
This study is a non randomized non comparative study with two Siddha formulations Sindhuvallathy Mezhugu and Kalladaippu Kudineer are available in Siddha classical texts existing for longer period. But there is no scientific data is documented about these formulations. This study aimed to evaluate the efficacy of the study drugs for urolithiasis. After the preliminary drug standardization the clinical study is Started at The National Institute of Siddha Tambaram. The primary outcome measure is either the Expulsion of stones or Changes in the number and size of the stones with 45 days drug treatment.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives. To assess the efficacy of sindhu vallathy mezhugu and Kalladaippu kudineer in Urolithiasis.

Secondary objectives

1. To standardize the study drugs.
2. To observe the adverse effects if any

Methods of proposed research:

The consists of two segments Part - A. Non- clinical studies -standardisation of the study drugs. Part - B. Clinical studies.

Study drugs

1. Sindhu Vallathy mezhugu will be prepared as per the literature Agasthiar vaidhya vallathy 600.
2. Kalldaippu Kudineer will be adapted from Athmaraktchamirtham Ennum Vaidhya Sarasangeeragam, 1968,page 349, 2.Siddha formulary of India part-II

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* both gender
* diagnosed ultrasonographically/radiographically with visible calculi of >5mm
* with or without clinical symptoms .

Exclusion Criteria:

* Patients with severe pain and not responding to pain killers
* Bilateral Calculi obstruction requiring immediate surgery,
* Existing renal failure,
* Pregnant and lactating women,
* Age<18 years,
* known hepatic and cardiac diseases,
* Subjects those who are not willing to give informed consent
* Women those who are planning for pregnancy .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Expulsion of stones or Reduction in the number and size of the stones. | 0,15,30,45 days post drug treatment
  The recruited subjects will be assessed for their parameters from base line and 15th day 30th day and 45th day of drug treatment. It will be measured either the expulsion of stones and/or reduction in number and size of stones from the baseline. The Ultra sound abdomen or X-ray will be done on 0 day and 45th day only.

SECONDARY OUTCOMES:
Prevention of stone forming factors within the study period. | 0,15th ,30th and 45th day
  All the clinical parameters and Investigatory parameters will be assessed from baseline and in every follow up visit till 45 days.
Reduction in pain and symptom score | 0 15 30 45 days
  Based on the reduction in the clinical symptoms
Changes in other investigations | 0 15th 30th 45th days
  Changes in other laboratory parameters lipid profile renal profile urinary parameters etc will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dr. K Rajalakshmi, M.D (s), Principal Investigator — The Tamilnadu Dr. MGR. Medical University
Locations (1):
- National Institute of Siddha, Chennai, Tamil Nadu, India